CLINICAL TRIAL: NCT05333029
Title: A Phase II Study of Combination Treatment with Extracorporeal Photopheresis and Mesenchymal Stem Cell Infusion for High-Risk and Steroid-Refractory Acute GVHD
Brief Title: Extracorporeal Photopheresis and Mesenchymal Stem Cell Infusion for GVHD
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Molly Gallogly (Other)
Responsible Party: Sponsor-Investigator, Molly Gallogly, Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE1Z20
Record Dates: First submitted 2022-04-04; First posted 2022-04-18 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-11

CONDITIONS: Graft Versus Host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — Photopheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- MSCs + ECP (Experimental): The treatment period consists of a single, 28-day cycle. Participants will be treated with ECP 2 to 3 times per week per the discretion of the treating physician. Participants will receive IV infusions of MSCs on days 1 (+ 2 days) and 8 (+/- 2 days). A third dose may be given on day 15 (+/- 2 days) if the principal investigator (PI) and treating physician determine the MSC infusions have benefited the participant.
  Participants will be followed for up to 1 year for assessment of endpoints.
  Interventions: Biological: Allogeneic mesenchymal stromal cells (MSCs); Biological: Extracorporeal photopheresis (ECP)

INTERVENTIONS:
Biological: Allogeneic mesenchymal stromal cells (MSCs) — Treatment dose 2 x10^6 cells/kg (+/- 20%)
Biological: Extracorporeal photopheresis (ECP) — Blood is collected through an intravenous (IV) line which is connected to an apheresis machine.The machine adds a chemical that makes the white blood cells sensitive to light. Then the machine shines a light on the cells and then returns the blood to the participant

SUMMARY:
The purpose of this study is to see if two treatments (extracorporeal photopheresis and Mesenchymal Stromal Cell (MSC) infusion, can be given safely together, and if they improve the symptoms of a Graft versus Host Disease (GvHD), a complication that can occur in people who undergo stem cell transplant.

DETAILED DESCRIPTION:
This is a Phase II study of human MSCs for the treatment of High-Risk aGVHD (HRaGVHD) and steroid-refractory acute GVHD (SRaGVHD). MSCs are cells that can help the body heal from injury and maintain a healthy immune system. MSCs have been used to prevent and treat a GvHD. In previous human studies, MSC infusion has been generally well-tolerated and safe, and in some cases, benefit was reported. The donor of the MSCs could be a relative or a stranger, and does not need to be the same individual who donated the stem cells for the stem cell transplant. All donors are screened for infectious diseases, similar to a blood donor. All donors have a physical exam.

Corticosteroids may be administered with MSCs/ECP. Continued use of anti-infective medications, GVHD prophylaxis medications (including calcineurin inhibitors), transfusion support, and topical steroid therapy is permitted. Participants will be assessed for safety and tolerability using a continuous monitoring approach. In order to be included in the tolerability review, participants must have received at least 1 treatment with MSCs.

ELIGIBILITY:
Inclusion Criteria:

-One of the following diagnoses:

--High risk aGVHD, either biopsy proven or clinical diagnosed as defined by either:

* Skin stage 4
* Lower gastrointestinal (GI) stage ≥ 3
* Liver stage ≥ 3
* Skin stage 3 and lower GI or liver stage ≥ 2 GVHD
* Hyper-acute GVHD as defined by aGVHD within the first 14 days of transplant
* Overall grade 2-4 aGVHD with high-risk disease identified by the Viracor Eurofins Symptomatic Onset or Post-Treatment Algorithm

OR:

--Steroid refractory aGVHD (either biopsy proven or clinical diagnosed) as defined by any one of the following criteria per NCCN (National Comprehensive Cancer Network) Guidelines for Hematopoietic Cell Transplantation (HCT):

* Progression of aGVHD within 3-5 days of therapy onset with ≥ 2 mg/kg/day of methylprednisolone or equivalent
* Failure to improve within 5-7 days of treatment initiation (2 mg/kg/day of methylprednisolone or equivalent)
* Incomplete response after more than 28 days of immunosuppressive treatment including steroids (2 mg/kg/day of methylprednisolone or equivalent)

  * Hct > 27 and plts > 50,000 x10^9/L (may be achieved via transfusion on ECP days)
  * Candidate for appropriate vascular access for ECP, which may include: (1) peripheral IV with 16 or 17 gauge Fistula needle; (2) central venous access device (apheresis catheter, tunneled central vascular access device), (3) vortex implanted port; (4) Bard POWERFLOW® implanted port
  * Eastern Cooperative Oncology Group Performance status ≤ 3
  * Participants who underwent an allogeneic hematopoietic stem cell transplantation from any donor source
  * Participants must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Active malignancy
* Contraindication to photopheresis, including any of the following: (1) known sensitivity to psoralen compounds such as 8-MOP; (2) comorbidities that may result in photosensitivity; (3) aphakia; (4) insufficient weight/circulating volume (defined by photopheresis machine characteristics); (5) hemodynamic instability; (6) platelet count < 20 x 109/μL despite platelet support; (7) bleeding diathesis; (8) hematocrit < 27 despite red blood cell support; (9) inability to lie flat for 4 hours; (10) inadequate venous access
* Participants with uncontrolled inter-current illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or breastfeeding women are excluded from this study because chemotherapy involved with RIC (Reduced-Intensity Conditioning) have the significant potential for teratogenic or abortifacient effects.
* Any condition that would, in the investigator's judgment, interfere with full participation in the study, including administration of study drug and attending required study visits; pose a significant risk to the participant; or interfere with interpretation of study data.
* Known allergies, hypersensitivity, or intolerance to any of the study medications, excipients, or similar compounds.
* Progressive underlying malignant disease or post-transplant lymphoproliferative disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Percent of participants with response to therapy | Day 28
  Response to therapy:
  Complete Remission (CR): Defined as the complete resolution of aGVHD symptoms in all organs, without secondary GVHD therapy.
  Partial Remission (PR): Defined as improvement in GVHD stage in all initial GVHD target organs without complete resolution and without worsening in any other GVHD target organs, without secondary GVHD therapy.
  The true response rate will be estimated based on the number of responses using a binomial distribution and its confidence interval will be estimated using Wilson's method

SECONDARY OUTCOMES:
aGVHD severity per Blood and Marrow Transplant Clinical Trials Network Manual of Operations (BMT MOP). | 100 days post-intervention
  Acute GVHD Staging per BMT MOP
  Stage 1:
  * Skin: Maculopapular Rash < 25% body surface area (BSA)
  * Gastrointestinal (GI): Diarrhea < 500 mL/day or persistent nausea
  * Liver: Total bilirubin 2.1-3 mg/dL
  Stage 2:
  * Skin: Maculopapular Rash 25-50% BSA
  * Gastrointestinal (GI): Diarrhea > 500 mL/day
  * Liver: Total bilirubin 3.1-6 mg/dL
  Stage 3:
  * Skin: Maculopapular Rash > 50% BSA
  * Gastrointestinal (GI): Diarrhea > 1000 mL/day
  * Liver: Total bilirubin 6.1-15 mg/dL
  Stage 4:
  * Skin: Generalized erythroderma with bullae
  * Gastrointestinal (GI): Diarrhea > 1500 mL/day
  * Liver: Total bilirubin >15 mg/dL
aGVHD incidence | 100 days post-intervention
  the number of participants that had acute GVHD incidence
Safety as measured by number of adverse events attributed to MSC and ECP therapy | Day 30
  To evaluate the total number of adverse events attributed to MSC and ECP therapy
Safety as measured by severity of adverse events attributed to MSC and ECP therapy | Day 30
  number of participants with adverse events (above or equal to grade 3) attributed to MSC and ECP therapy
Number of participants with non-relapse mortality (NRM) | 1 year
Number of participants with relapse-related mortality | 1 year
Average time to relapse | 1 year
  Average time to relapse. The Kaplan-Meier method will be used to estimate survivor function
Chronic GVHD incidence | At 1 year from the start of treatment
  the number of participants that had Chronic GVHD incidence
Overall Survival (OS) | 1 year
  Average OS. The Kaplan-Meier method will be used to estimate survivor function
Steroid dose decrease | Up to day 28
  change in steroid dose from day 1 to day 28
Steroid discontinuation rate | Up to day 28
  Percentage of patients who are no longer taking systemic corticosteroids at day 28
Change in FACT-BMT (Functional Assesment of Cancer Therapy-Bone Marrow Transplant) survey score | 1 year
  Quality of life survey scores measured by change in FACT-BMT survey scores. The Functional Assessment of Cancer Therapy-General (FACT-G) subscales, total score on their 12-item BMT subscale including physical, social, emotional and functional well-being measured over time will be summarized by mean and standard deviation at each time point.
  The QOL data will be further analyzed using repeated measures regression models, i.e., mixed-effects models 28-30 ,28-30 with an unstructured covariance matrix and a categorical effect of time to calculate between-group differences in improvement from baseline in these QOL outcomes
Percent regulatory T cells (% Tregs) | Up to 1 year after treatment
  T cell subsets in responders vs. nonresponders as measured by percent Tregs
CD4:CD8 ratio | Up to 1 year after treatment
  T cell subsets in responders vs. nonresponders as measured by cluster of differentiation (CD)4:CD8 ratio

CONTACTS AND LOCATIONS:
Overall Officials: Molly Gallogly, MD, PhD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie or influence the results observed from the study
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Beginning 3 months and ending 5 years following article publication
Access Criteria: Investigators who provide a methodologically sound proposal for use of requested data